CLINICAL TRIAL: NCT05910281
Title: Rebound Pain and Related Factors in Patients Who Underwent Femoral Nerve Block for Postoperative Pain Control in Total Knee Arthroplasty
Brief Title: Rebound Pain and Related Factors in Postoperative Patients With Total Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Bilal Katipoglu, M.D, Gulhane Training and Research Hospital
Other Study IDs: E2-23-4135
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Pain; Postoperative Complications; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications; Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this prospective observational study is to detect rebound pain and related factors in postoperative patients with total knee arthroplasty.

DETAILED DESCRIPTION:
Total knee arthroplasty is an effective treatment method for knee osteoarthritis and because it is an invasive method, more than 50% of patients experience postoperative pain. Peripheral nerve blocks are widely used for optimal pain control. The femoral block is a frequently preferred peripheral nerve block method for postoperative analgesia in total knee arthroplasty surgery. However, after peripheral nerve block, a condition called rebound pain (rebound pain), which is described as very severe pain, lasting about 2 hours, usually of the burning type, occurs. The aim of this prospective observational study is to detect rebound pain and related factors in postoperative patients with total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years older age who underwent total knee arthroplasty

Exclusion Criteria:

* ASA score 4 or >4
* Active infection
* End stage organ failure
* Pregnancy
* Established diagnosis neuropsychiatric disease ( epilepsy, neuropathy, neuromuscular disease, cerebrovascular disease...)
* Uses of oral corticosteroids

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - 18-80 years older age who underwent total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | postoperative 3-5 days fellow-up
  The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, None Selected, Turkey (Türkiye)